CLINICAL TRIAL: NCT04287530
Title: Poly-unsaturated Fatty Acids and Developmental Dyslexia: Correlations With Cognitive Performance and Effects of Supplementation in Addition to Neuropsychological Treatment
Brief Title: Poly-unsaturated Fatty Acids and Developmental Dyslexia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: University of Milan (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 677
Record Dates: First submitted 2020-02-20; First posted 2020-02-27 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Dyslexia, Developmental
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tachidino + PUFA supplementation (Experimental): Group 1 will be treated with the usual rehabilitation protocol adopted at IRCCS E. Medea (remote intervention delivered through the Tachidino platform). The program will be delivered during four weeks, starting two months after the pre-testing session. Additionally, the children will receive daily supplementation with 6 daily PUFA (Omega-3 and Omega-6) chewable capsules from the beginning (immediately after the pre-testing session) to the end (immediately before the post-testing session) of the observation period, for a total of three months.
  Interventions: Dietary Supplement: Poly-unsaturated fatty acids supplementation; Behavioral: Neuropsychological intervention
- Tachidino + Placebo (Active Comparator): Group 2 will be treated with the usual rehabilitation protocol adopted at IRCCS E. Medea (remote intervention delivered through the Tachidino platform), delivered during four weeks, starting two months after the pre-testing session, exactly as Group 1. Additionally, the children will receive daily supplementation with 6 daily Placebo (triglycerides) chewable capsules from the beginning (immediately after the pre-testing session) to the end (immediately before the post-testing session) of the observation period, for a total of three months.
  Interventions: Behavioral: Neuropsychological intervention; Dietary Supplement: Placebo
- PUFA supplementation (Experimental): Groups 3 will receive only daily supplementation with 6 daily PUFA (Omega-3 and Omega-6) chewable capsules from the beginning (immediately after the pre-testing session) to the end (immediately before the post-testing session) of the observation period, for a total of three months.
  Interventions: Dietary Supplement: Poly-unsaturated fatty acids supplementation
- Placebo (Placebo Comparator): Groups 4 will receive only daily supplementation with 6 daily Placebo (triglycerides) chewable capsules from the beginning (immediately after the pre-testing session) to the end (immediately before the post-testing session) of the observation period, for a total of three months.
  Interventions: Dietary Supplement: Placebo
- Control group (No Intervention): Typically Developing participants, as a comparison group for experimental tasks and for PUFA levels in the blood

INTERVENTIONS:
Dietary Supplement: Poly-unsaturated fatty acids supplementation — Daily supplementation with 6 daily PUFA (Omega-3 and Omega-6) chewable capsules from the beginning (immediately after the pre-testing session) to the end (immediately before the post-testing session) of the observation period, for a total of three months.
  Other Names: Equazen Eye Q chewable capsules
  Arms: PUFA supplementation; Tachidino + PUFA supplementation
Behavioral: Neuropsychological intervention — Rehabilitation protocol adopted at IRCCS "E. Medea" (remote intervention delivered through the Tachidino platform), delivered during four weeks, starting two months after the pre-testing session.
  Other Names: Tachidino
  Arms: Tachidino + PUFA supplementation; Tachidino + Placebo
Dietary Supplement: Placebo — Daily supplementation with 6 daily Placebo (triglycerides) chewable capsules from the beginning (immediately after the pre-testing session) to the end (immediately before the post-testing session) of the observation period, for a total of three months.
  Other Names: Equazen Eye Q red Placebo chewable capsules
  Arms: Placebo; Tachidino + Placebo

SUMMARY:
Poly-unsaturated fatty acids (PUFAs) represent a component of lipids that covers a relevant role in human diet and biological functions such as provision of energy, functionality of cell membranes and tissue metabolism. Fatty acids carbon chains can be saturated (with no presence of double bonds) or unsaturated (with one or more double bonds). PUFAs fall into the unsaturated group, and they can be divided into two classes: omega-3 (n-3) and omega-6 (n-6) fatty acids (FAs). PUFAs are relevant components of cellular membranes, phospholipids, and precursors of eicosanoids, which influence neuronal development and functioning, docosahexaenoic acid (DHA) and arachidonic acid (AA) in fact are involved in cell growth, neural signaling, and gene expression. The main natural dietary source for Eicosapentaenoic acid (EPA) and DHA is fish oil. It has also been shown how the Magnocellular system, which includes the retinal ganglion cells, the lateral geniculate nucleus (for the visual system, while the medial geniculate nucleus would be involved for the auditory system) of the thalamus, the posterior parietal cortex, various areas visual of the cortex and part of the cerebellum, is sensitive to the contribution of fatty acids through nutrition. A deficit related to the Magnocellular system, specialized in the processing of stimuli with high temporal frequencies and low spatial frequencies, in both the visual and auditory modalities, has been proposed as one of the causes of Developmental Dyslexia (DD). According to this hypothesis, an alteration at the magnocellular level would affect reading by hampering temporal processing of the visual signal and would reduce the quality of the phonological representations due to imperfect acoustic analysis of the incoming phonemes. It is therefore possible to hypothesize that supplementation of PUFA in dyslexic children would improve the functions of the M-system and thus create better conditions to the remediation of reading difficulties, especially through remediation programs specifically tapping visual attention and rapid processing of visual stimuli. The remediation program currently used at Scientific Institute (IRCCS) Medea, "Tachidino", based on tachistoscopic, hemisphere-specific stimulation and on training of selective visual-spatial attention, has exactly these characteristics.

Hence, the present study aims to test the efficacy of PUFA supplementation before and during treatment with Tachidino.

ELIGIBILITY:
Inclusion Criteria for DD participants will be:

* A formal diagnosis of Developmental Dyslexia, Specific Reading Disorders or Mixed Learning Disorders
* Age between 7 and 15
* Attending at least the third class of primary school
* Monolingual speakers or bilingual speakers with perfect mastery of the Italian language (equivalent to monolinguals)
* Intelligence Quotient (IQ) >= 80
* At least one z-score below -2 Standard Deviations from age mean in at least one of the following tests: text reading, word reading, nonword reading (Dyslexia and Dysorthography (DDE-2) battery, Memory Training (MT) tests)
* Not having received any specific rehabilitation treatment for dyslexia before

Inclusion criteria for control participants will be:

* Age between 7 and 15
* Attending at least the third class of primary school
* Monolingual speakers or bilingual speakers with perfect mastery of the Italian language (equivalent to monolinguals)
* no reported record of difficulties with reading nor specific learning disorders
* Intelligence Quotient (IQ) >= 80
* No z-score below -1,5 Standard Deviations from age mean in any of the following tests: text reading, word reading, nonword reading ("DDE-2" battery, "MT" tests)

Exclusion Criteria:

* Intellectual disability
* Attention Deficit with Hyperactivity (ADHD)
* Neurological disorders
* Sensory deficits that are not /cannot be corrected-to-normal by lenses or hearing aids.
* Allergy to fish and shellfish
* Absorption Disorders (malabsorption)
* Children already (or recently) on a diet with PUFA supplementation
* Children on a therapy with psychoactive medications (anti-depressant, anxiety-control etc.) or with supplements who have not reached a stable administration schedule.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2020-05-02 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
PUFA supplementation effects on the results of neuropsychological intervention | 3 months
  Difference in treatment-related changes (post-test minus pre-test) observed in reading measures (speed and accuracy in word, nonword and text reading; average of the scores expressed as z-scores with respect to age norms) between the experimental group (Tachidino + PUFA supplementation) and the comparison group (Tachidino + placebo)

SECONDARY OUTCOMES:
Changes in Rapid Automatized Naming (RAN) due to supplementation with PUFAs | 3 months
  Difference in change-scores (i.e. post-test minus pre-test) observed in Rapid Automatized Naming (z-scores with respect to age norms) in the experimental group versus placebo
Changes in visual search functions due to supplementation with PUFAs | 3 months
  Difference in change-scores (i.e. post-test minus pre-test) observed in Visual Search scores (z-scores with respect to age norms) in the experimental group versus placebo
Changes in Magnocellular functions due to supplementation with PUFAs | 3 months
  Difference in change-scores (i.e. post-test minus pre.test scores) observed in neuropsychological measures related to Magnocellular functions (Magnocellular tasks in the visual modality, efficiency expressed in msec) in the experimental group versus placebo
Correlations between blood levels of PUFA and reading performance | Baseline
  Pearson's correlation index between PUFA levels in the blood (Ratio omega-6/omega-3) and reading performance expressed in z-scores
Correlations between blood levels of PUFA and writing performance | Baseline
  Pearson's correlation index between PUFA levels in the blood (Ratio omega-6/omega-3) and writing performance expressed in z-scores
Change in blood levels of PUFAs in children with Dyslexia | 3 months
  Changes (post-test versus pre-test levels) in blood levels of PUFAs (Ratio omega-6/omega-3) for children with DD after 3 months supplementation
Changes in blood levels of PUFAs relate to changes in reading performance in children with Dyslexia | 3 months
  Pearson's correlation index between changes in PUFA levels (i.e. post-test minus pre-test levels) in the blood (Ratio omega-6/omega-3) and change-scores (i.e. post-test minus pre-test scores) in reading performance in children with DD (expressed in z-scores)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Lorusso, PhD, Principal Investigator — IRCCS Eugenio Medea
Locations (2):
- Italy (2):
  - IRCCS "E. Medea" - La Nostra Famiglia, Bosisio Parini, (LC)
  - IRCCS E.Medea, polo di Conegliano, Conegliano, TV

REFERENCES:
- [Background] Borasio F, Syren ML, Turolo S, Agostoni C, Molteni M, Antonietti A, Lorusso ML. Direct and Indirect Effects of Blood Levels of Omega-3 and Omega-6 Fatty Acids on Reading and Writing (Dis)Abilities. Brain Sci. 2022 Jan 27;12(2):169. doi: 10.3390/brainsci12020169. PMID 35203933
- [Background] Borasio F, De Cosmi V, D'Oria V, Scaglioni S, Syren ME, Turolo S, Agostoni C, Coniglio M, Molteni M, Antonietti A, Lorusso ML. Associations between Dietary Intake, Blood Levels of Omega-3 and Omega-6 Fatty Acids and Reading Abilities in Children. Biomolecules. 2023 Feb 15;13(2):368. doi: 10.3390/biom13020368. PMID 36830737